CLINICAL TRIAL: NCT00433004
Title: A Pilot Randomized Control Trial of Advanced Supply of Levonorgestrel Emergency Contraception vs. Routine Postpartum Contraceptive Care in the Teenage Population
Brief Title: Advance Supply of Emergency Contraception Compared to Routine Postpartum Care in Teens
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 805358
Record Dates: First submitted 2007-02-08; First posted 2007-02-09 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Post Partum
Keywords: Teen; Plan B; Post Partum; Emergency Contraception
MeSH Terms: interventions — Levonorgestrel

ARMS (2):
- 1 (No Intervention): No advance supply of emergency contraception
- 2 (Active Comparator): Advance supply of emergency contraception is given
  Interventions: Drug: Plan B (Levonorgestrel)

INTERVENTIONS:
Drug: Plan B (Levonorgestrel) — PP TEENS ARE RANDOMIZED TO PLAN B + ROUTINE CONTRACETIVE CARE VS. ROUTINE CARE ALONE. QUESTIONNAIRES ON HEALTH STATUS, SEXUAL HISTORY, AND CONTRACEPTIVE USE ARE COMPLETED AT STATED INTERVALS.
  Arms: 2

SUMMARY:
This is a pilot randomized controlled trial to assess the effects of advanced supply of emergency contraception versus routine care in a teen postpartum population. The goals are to assess feasibility of recruiting and retaining postpartum teens; to obtain estimates of the prevalence of (use of Plan B, primary contraceptive continuation, unprotected intercourse exposure, and pregnancy rates), in postpartum teens given advanced supply of Plan B; to assess whether or not (lack of use of Plan B, contraceptive method non-continuation, and unprotected intercourse exposure), are surrogate markers for risk of unintended pregnancy.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. English speaking
3. Aged 14-19 at enrollment
4. Immediately postpartum of a live infant
5. Planning to parent the baby
6. Desiring to delay another pregnancy for at least one year
7. General good health
8. Willing and able to follow the study protocol

Exclusion Criteria

1. Allergy to levonorgestrel
2. Current substance abuse
3. Plans for relocation outside of Philadelphia

Ages: 14 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Schreiber, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Advance EC: No advance supply of emergency contraception
- Advance EC Given: Advance supply of emergency contraception is given
  Plan B (Levonorgestrel): PP TEENS ARE RANDOMIZED TO PLAN B + ROUTINE CONTRACETIVE CARE VS. ROUTINE CARE ALONE. QUESTIONNAIRES ON HEALTH STATUS, SEXUAL HISTORY, AND CONTRACEPTIVE USE ARE COMPLETED AT STATED INTERVALS.
Period: Overall Study
Arm/Group | No Advance EC | Advance EC Given
Started | 27 | 23
Completed | 22 | 16
Not Completed | 5 | 7
Not completed — Lost to Follow-up | 5 | 7

BASELINE CHARACTERISTICS:
Groups:
- Advance EC Given: Advance supply of emergency contraception is given
  Plan B (Levonorgestrel): Postpartum TEENS ARE RANDOMIZED TO PLAN B + ROUTINE CONTRAPCETIVE CARE VS. ROUTINE CARE ALONE. QUESTIONNAIRES ON HEALTH STATUS, SEXUAL HISTORY, AND CONTRACEPTIVE USE ARE COMPLETED AT STATED INTERVALS.
- Total: Total of all reporting groups
Arm/Group | No Advance EC | Advance EC Given | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Continuous [Mean (Full Range); unit: years] | 17.6 [14 to 19] | 17.6 [14 to 19] | 17.6 [14 to 19]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: ABILITY TO FOLLOW POSTPARTUM TEENS FOR 1 YEAR.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | No Advance EC | Advance EC Given
Number analyzed (Participants) | 27 | 23
Participants | 22 | 16

2. Primary Outcome: PREGNANCY RATES
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | No Advance EC | Advance EC Given
Number analyzed (Participants) | 27 | 23
Participants | 8 | 3

3. Primary Outcome: PLAN B USE
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | No Advance EC | Advance EC Given
Number analyzed (Participants) | 27 | 23
Participants | 8 | 12

ADVERSE EVENTS:
Arm/Group | No Advance EC | Advance EC Given
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No